CLINICAL TRIAL: NCT01269931
Title: Evaluation of Clinical Endobronchial Ultrasound Skills Following Clinical Versus Simulation Training.
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: David Ryan Stather, University of Calgary
Other Study IDs: E-23051
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-12

CONDITIONS: EBUS-TBNA Training Methods
Keywords: endobronchial ultrasound; bronchoscopy; education; interventional bronchoscopy; simulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1 (EBUS-TBNA simulator training): Group 1 (EBUS-TBNA simulator training): pulmonary medicine trainees with >30 bronchoscopy procedures experience, >nine months of pulmonary fellowship training and no clinical EBUS-TBNA experience (n=4).
  Interventions: Procedure: EBUS-TBNA
- Group 2 (Clinical EBUS-TBNA training): Group 2 (Clinical EBUS-TBNA training): pulmonary medicine trainees in the 2nd half of their final year of pulmonary training or recent graduates (within one year), with >50 bronchoscopy procedures experience who completed a one-month elective with the Interventional Pulmonary Medicine (IPM) service with ≥15 and ≤25 EBUS-TBNA procedures experience (n=4).
  Interventions: Procedure: EBUS-TBNA

INTERVENTIONS:
Procedure: EBUS-TBNA — Endobronchial ultrasound with transbronchial needle aspiration (EBUS-TBNA) is a revolutionary diagnostic pulmonary procedure that allows visualization and safe, accurate biopsies of intra-thoracic structures during bronchoscopy. Patients enrolled in this study at the University of Calgary would have undergone this procedure regardless of being enrolled in this study. The purpose of the study was to prospectively compare the EBUS-TBNA performance of 2 groups of learners, performing EBUS-TBNA on patients, who had received to different methods of EBUS-TBNA training. Patients were randomly assigned to undergo bronchoscopy with a trainee from Group 1 or Group 2.
  Other Names: - endobronchial ultrasound; - EBUS

SUMMARY:
Bronchoscopy is a procedure whereby a small flexible camera is used to inspect and biopsy abnormalities in the lungs. Linear endobronchial ultrasound with transbronchial needle aspiration (EBUS-TBNA) is a revolutionary diagnostic pulmonary procedure that allows visualization and safe, accurate biopsies of structures in and around the lungs during bronchoscopy. EBUS-TBNA can be challenging to learn.

Historically, bronchoscopy has been taught using an apprenticeship model, whereby trainees practice on patients. With the introduction of computer bronchoscopy simulators, trainees can now obtain basic bronchoscopy skills by practicing on the simulator, rather than practicing on patients.

This study aims to compare trainee EBUS-TBNA performance during actual procedures on patients, following training with a computer EBUS-TBNA simulator versus conventional clinical EBUS-TBNA training (trainees taught by practicing on patients). Our hypothesis is that the skills learned using a computer EBUS-TBNA simulator are transferable to clinical EBUS-TBNA performance, meaning that using a computer EBUS-TBNA simulator for training is just as good as learning these skills by practicing on patients.

The use of EBUS-TBNA simulators for training could have the advantage of minimizing the burden of procedural learning on patients.

DETAILED DESCRIPTION:
Learners in Group 1 undergo training on the EBUS-TBNA simulator before performing EBUS-TBNA on the study patients.

Learners in Group 2 completed a one month clinical Interventional Pulmonary Medicine rotation. During this rotation, they completed ≥15 and ≤25 EBUS-TBNA clinical procedures with an Interventional Pulmonologist experienced in EBUS-TBNA.

Learners in both groups receive a standard EBUS-TBNA knowledge review process before their patient care EBUS-TBNA experience. This includes a series of oral questions and a written lymph node staging diagram which they need to correctly answer, prior to performing EBUS-TBNA on study patients. Learners in Group 2 complete this review process informally on a number of occasions during their Interventional Pulmonary Medicine rotations. Learners in Group 1 formally undergo this review process 5 times during the EBUS-TBNA simulation training.

Bronchoscopy is performed utilizing a 1T-160 Olympus video bronchoscope (Olympus Canada, Markham, Canada) for the airway examination and a BF-UC160F-OL8 (EBUS bronchoscope - Olympus Canada, Markham, Canada) for the EBUS-TBNA procedure. In order to standardize for differences in bronchoscopy method, a single attending Interventional Pulmonologist (IP) is responsible for performing all 16 bronchoscopies with the learners. The complete airway examination and any additional non-EBUS-TBNA samples are performed by the attending IP. All endobronchial ultrasound bronchoscopy performance metrics are recorded by another IP not involved in the procedure on a standard data sheet.

EBUS-TBNA is performed by the learner with 3 specific goals:

1. Intubation with the EBUS-TBNA bronchoscope.
2. Lymph Node Ultrasound Examination. Identify 5 major lymph node stations (11R, 4R, 7, 4L, 11L).
3. Sampling of two lymph nodes per patient. The order and location of lymph nodes was at the discretion of the attending IP. Following the biopsy of two lymph nodes stations by the learner, the attending IP completes the rest of the procedure, including any further biopsies that are necessary. The learner is expected to perform 3 successful passes in each of the two lymph nodes, with a total of 5 allowed attempts per lymph node station.

The learner procedure time starts at the time of the first intubation attempt with the EBUS-TBNA bronchoscope, and finishes with the last biopsy of the second lymph node station. If other clinically important lymph nodes are present or if more than 3 successful aspirations are desired, the stopwatch is stopped while the attending IP performed the biopsies.

Samples are placed in alcohol preservative and sent to the cytopathology lab as per our routine procedure. No indication as to group allocation is available to the clinical cytopathologist interpreting the samples.

To be enrolled, patients and learners must give written informed consent.

The EBUS-TBNA simulator used for this study is the AccuTouch Flexible Bronchoscopy Simulator (CAE Healthcare, Montreal, Canada), equipped with an EBUS-TBNA module. This simulator has been described in detail previously in the articles cited at the end of this ClinicalTrials.gov entry.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* suspected lung cancer patients with mediastinal adenopathy
* at least 2 enlarged mediastinal or hilar lymph nodes (one >1.0 cm and one >1.5 cm in short axis on CT Chest, one of the lymph nodes must be in position 7 or 4R
* eighteen years of age or older

Exclusion Criteria:

* Lack of informed consent
* any contraindication to bronchoscopy
* any significant severe co-morbidities (i.e. severe obstructive lung disease, active cardiac disease such as angina)

Learners:

Group 1 (EBUS-TBNA simulator training):

Inclusion Criteria:

* pulmonary medicine trainees with >30 bronchoscopy procedures experience, >nine months of pulmonary fellowship training and no clinical EBUS-TBNA experience (n=4)

Exclusion Criteria:

* lack of informed consent

Group 2 (Clinical EBUS-TBNA training):

Inclusion Criteria:

* pulmonary medicine trainees in the 2nd half of their final year of pulmonary training or recent graduates (within one year), with >50 bronchoscopy procedures experience who completed a one-month elective with the Interventional Pulmonary Medicine (IPM) service with ≥15 and ≤25 EBUS-TBNA procedures experience (n=4).

Exclusion Criteria:

* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective, comparative study of 2 groups of learners, performing EBUS-TBNA on patients. Patients are randomly assigned to undergo bronchoscopy with a trainee from Group 1 or Group 2. Learners are pulmonary medicine trainees at the University of Calgary. Patients are suspected lung cancer patients with mediastinal adenopathy seen by the University of Calgary Interventional Pulmonary Medicine service.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
total learner EBUS-TBNA procedure time/number of successful aspirations | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure

SECONDARY OUTCOMES:
total learner EBUS-TBNA procedure time | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
time to intubation | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
lymph node ultrasound examination time | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
percentage of successful aspirations | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
number of intubation attempts | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
percentage of lymph node stations correctly identified during lymph node ultrasound examination | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
number of instructional comments required by the attending pulmonologist | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
sample adequacy | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
diagnostic yield | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
expert respiratory therapist subjective EBUS-TBNA technical skill assessment | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
total lymph node biopsy time | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
time to EBUS-TBNA intubation | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
number of unsuccessful biopsies per case | patients followed for 2 months or until death - measured at patient EBUS-TBNA procedure
  includes a list of reasons for unsuccessful biopsies: bronchoscope damage, contaminated sample, penetrating far side of lymph node, missing the lymph node, vascular puncture

CONTACTS AND LOCATIONS:
Overall Officials: David R Stather, MD, Principal Investigator — University of Calgary
Locations (1):
- Dr. David R Stather, Calgary, Alberta, Canada

REFERENCES:
- [Result] Stather DR, Maceachern P, Rimmer K, Hergott CA, Tremblay A. Validation of an endobronchial ultrasound simulator: differentiating operator skill level. Respiration. 2011;81(4):325-32. doi: 10.1159/000323520. Epub 2011 Feb 9. PMID 21311171
- [Result] Stather DR, MacEachern P, Rimmer K, Tremblay A. Assessment of Endobronchial Ultrasound Skills Following Clinical vs Simulator Training. Chest 2010;138:589A
- See also: Website for the University of Calgary Interventional Pulmonary Medicine Program — http://ucalgary.ca/ipm